CLINICAL TRIAL: NCT03764085
Title: Open-label, Randomized, Controlled, With Blind Assessor, Study to Assess Efficacy and Safety of Rheosorbilact®, Solution for Infusion, in Comparison With Ringer's Lactate, Solution for Infusion, in a Complex Therapy of Sepsis.
Brief Title: Efficacy and Safety of Rheosorbilact® Solution for Infusion, in a Complex Therapy of Sepsis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuria-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RheoSTAT-CP0620
Record Dates: First submitted 2017-10-10; First posted 2018-12-04 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-01

CONDITIONS: Sepsis; Intoxication; Septic
MeSH Terms: conditions — Sepsis; Toxemia | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will perform the assessment of primary, secondary efficasy and safety parameters
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheosorbilact® (Experimental): Rheosorbilact® is administered as a part of the infusion therapy intravenously (with speed 40-60 drip per minute) at a dose of 600 to 1,000 ml (10 to 15 ml/kg body weight per 24 hours).The period of the treatment with the study drug lasts 3 days.
  Interventions: Drug: Rheosorbilact®
- Ringer's Lactate (Active Comparator): Ringer's Lactate is administered as a part of the infusion therapy intravenously (with speed 40-60 drip per minute) at a dose of 1,000 to 2,500 ml (15 to 40 ml/kg body weight per 24 hours).The period of the treatment with the active comparator lasts 3 days.
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Rheosorbilact® — Administered intravenously (with speed 40-60 drip per minute) at a dose of 600 to 1,000 ml (10 to 15 ml/kg body weight per 24 hours) for 3 days.
  Arms: Rheosorbilact®
Drug: Ringer lactate — Administered intravenously (with speed 40-60 drip per minute) at a dose of 1,000 to 2,500 ml (15 to 40 ml/kg body weight per 24 hours) for 3 days.
  Arms: Ringer's Lactate

SUMMARY:
This study evaluates the efficacy and safety of Rheosorbilact®, solution for infusion ("Yuria-Pharm" LLC), in comparison with Ringer's Lactate, solution for infusion, in a complex therapy of sepsis. Half of participants will receive Rheosorbilact® in complex therapy, while the other half will receive Ringer's Lactate in complex therapy.

DETAILED DESCRIPTION:
Rheosorbilact® has rheological, anti-shock, detoxification, and alkalizing effects. Sorbitol and sodium lactate are the major pharmacologically active ingredients. In the liver, sorbitol is first converted into fructose, which is then converted into glucose, and then into glycogen. Part of sorbitol is used for urgent energy needs, while the other part is kept as a reserve in the form of glycogen. Isotonic sorbitol solution has a disaggregating effect and, therefore, improves microcirculation and tissue perfusion.

The management of metabolic acidosis with sodium lactate goes more slowly compared to bicarbonate solution, as far as sodium lactate enters the metabolic process; however the latter does not cause swings in pH values. The effect of sodium lactate is typically seen 20 to 30 minutes after administration.

Sodium chloride is a plasma-substituting agent that exhibits a detoxification and rehydration effect. It replenishes the deficiency of sodium and chlorine ions in various pathological conditions.

Calcium chloride replenishes deficiency of calcium ions. Calcium ions are essential in the transmission of nerve impulses, contraction of skeletal and smooth muscles, myocardial activity, bone tissue formation, and blood clotting. It reduces the permeability of cells and vascular walls, prevents the development of inflammatory reactions, enhances the resistance of the body to infections and can significantly boost phagocytosis.

Potassium chloride restores the water-electrolyte balance. It exhibits a negative chrono- and bathmotropic action and, when administered in high doses, has a negative ino- and dromotropic and moderate diuretic effect. It is involved in the process of nerve impulse conduction, increases the content of acetylcholine and causes excitation of the sympathetic segment of the autonomic nervous system and improves the contraction of skeletal muscles in subjects with muscular dystrophy or myasthenia.

Rheosorbilact® is administered to improve capillary blood flow for the prevention and treatment of traumatic, surgical, hemolytic, toxic and burn shock, acute blood loss, and burn disease; infectious diseases accompanied by intoxication, exacerbation of chronic hepatitis; sepsis, pre- and postoperative period to improve arterial and venous circulation for the prevention and treatment of thrombosis, thrombophlebitis, endarteritis, and Raynaud's disease.

Ringer's Lactate, solution for infusion will be used as a comparator. As a rehydrating agent, Ringer's Lactate has a detoxification effect, replenishes the deficiency of circulating blood volume, and stabilizes the water and electrolyte composition of blood. Ringer's Lactate normalizes the acid-base balance. Lactate is metabolized in the body to bicarbonate, so the solution has an alkalizing effect. With osmolarity at 273 mOsm/l, Ringer's Lactate is close to isotonic solution and is indicated for hypovolemia, isotonic dehydration, and metabolic alkalosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 to 60 years inclusive
2. Sepsis diagnosed according to ACCP / SCCM criteria (no later than 24 hours from the time of diagnosis of sepsis to screening visit) (Annex 1: Sequence Diagnostic Criteria for SCCM / ESICM / ACCP / ATS / SIS)
3. Informed consent for participation in the study signed by subject's own hand.
4. The baseline value of the SOFA scale ≥ 2 points.

Non-inclusion Criteria:

1. The presence of any of the criteria for severe sepsis by ACCP / SCCM (presence of signs of organ failure - Annex 1: criteria for diagnosis of sepsis SCCM / ESICM / ACCP / ATS / SIS)
2. Individual intolerance of the components of the study drug and the comparator;
3. Hypersensitivity to sodium lactate;
4. Intravenous infusions of lactate- or sorbitol-containing products within 24 hours before enrollment;
5. Pregnancy or breast-feeding;
6. Severe renal dysfunction (creatinine is more than 300 μmol/l or estimated creatinine clearance is less than 30 ml/min);
7. Metabolic alkalosis;
8. Severe metabolic acidosis;
9. Intracerebral hemorrhage;
10. Any thromboembolism;
11. Decompensated cardiovascular failure;
12. Arterial hypertension III st;
13. Conditions associated with immunodeficiency (the use of cytostatics or system steroids, AIDS);
14. Extracellular hyperhydration or hypervolemia;
15. Severe renal insuffiency (with oliguria / anuria);
16. Hyperkalaemia;
17. Hypercalcemia;
18. Ascites associated with cirrhosis;
19. Conditions associated with increased lactate levels (hyperlactatemia > 2 mmol / l), including lactic acidosis, or impaired lactate uptake (including due severe hepatic insufficiency);
20. Concomitant therapy with cardiac glycosides;

Exclusion Criteria:

1. Infusion of the study drug or the comparator is started more than 12 hours after randomization;
2. Lack of data for sepsis (diagnosis not confirmed);
3. Withdrawal of the informed consent by the subject;
4. Investigator considers that the infusion therapy with either study drug or comparator may not be continued for safety reasons;
5. Development of conditions that prevent further use of the study drug/comparator before efficacy evaluation visit (Visit 3);
6. Subject needs concomitant therapy prohibited in the study before efficacy evaluation visit (Visit 3);
7. Development of conditions (including serious adverse events) which make it impossible to evaluate the primary endpoint;
8. Confirmation of pregnancy at any time of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
A change in the total SOFA score vs. baseline score upon admission; | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Sequential Organ Failure Assessment (SOFA) score is composed of scores of six organ systems: R-respiratory, C-cardiovascular, H-hepatic, Co-coagulation, Re-renal, and N-neurological graded from 0 to 4 according to the degree of dysfunction or failure.
  The SOFA score ranges from 0 to 24 points. We evaluate initial SOFA score and differences between subsequent scores (Δ-SOFA scores).

SECONDARY OUTCOMES:
A change in the total APACHE II score vs. baseline score upon admission; | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Acute physiology and chronic health evaluation（APACHE) II score is calculated from a patient's age (0-6 points) and 12 physiological parameters (each item 0-4 points): AaDO2 or PaO2 (depending on FiO2), Temperature (rectal), Mean arterial pressure, pH arterial, Heart rate, Respiratory rate, Sodium (serum), Potassium (serum), Creatinine, Hematocrit, White blood cell count, Glasgow Coma Scale and chronic disease health status (0-5 points).
  The APACHE II score ranges from 0 to 71 points. We evaluate initial APACHE II score and differences between subsequent scores (Δ-APACHE II scores).
A change in the total SAPS II score vs. baseline score upon admission | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  The SAPS II score is made of 17 variables: 12 physiology variables, age, type of admission (scheduled surgical, unscheduled surgical, or medical), and three underlying disease variables (acquired immunodeficiency syndrome, metastatic cancer, and hematologic malignancy).
  The SAPS II score ranges from 0 to 160 points. We evaluate initial SAPS II score and differences between subsequent scores (Δ-SAPS II scores).
A change in the total MODS score vs. baseline score upon admission | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  MODS (Multiple Organ Dysfunction Score) is composed of scores of six organ systems: R-respiratory, C-cardiovascular, H-hepatic, Co-coagulation, Re-renal, and N-neurological graded from 0 to 4 according to the degree of dysfunction or failure.
  The MODS score ranges from 0 to 24 points. We evaluate initial MODS score and differences between subsequent scores (MODS scores).
Concentration of glucose | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of glucose (mmol/L) in blood serum after 8-hour fasting.
Concentration of sodium | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of sodium (mmol/L) in blood serum after 8-hour fasting.
Concentration of potassium | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of potassium (mmol/L) in blood serum after 8-hour fasting.
Concentration of lactate | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of lactate (mmol/L) in blood serum after 8-hour fasting.
Concentration of pyruvate | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of pyruvate (mmol/L) in blood serum after 8-hour fasting.
Concentration of urea | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of urea (mmol/L) in blood serum after 8-hour fasting.
Concentration of creatinine | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of creatinine (µmol/L) in blood serum after 8-hour fasting.
Concentration of bilirubin | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of bilirubin (µmol/L) in blood serum after 8-hour fasting.
Concentration of alanine aminotransferase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of alanine aminotransferase (U/L) in blood serum after 8-hour fasting.
Concentration of aspartate aminotransferase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of aspartate aminotransferase (U/L) in blood serum after 8-hour fasting.
Concentration of lactate dehydrogenase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of lactate dehydrogenase (U/L) in blood serum after 8-hour fasting.
Concentration of alkaline phosphatase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of alkaline phosphatase (U/L) in blood serum after 8-hour fasting.
Concentration of creatine kinase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of creatine kinase (U/L) in blood serum after 8-hour fasting.
Concentration of γ-Glutamyltransferase | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of γ-Glutamyltransferase (U/L) in blood serum after 8-hour fasting.
Concentration of low-molecular-weight adiponectin (LMW) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of low-molecular-weight adiponectin (U/L) in blood serum after 8-hour fasting.
Concentration of middle-molecular-weight adiponectin (MMW) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of middle-molecular-weight adiponectin (U/L) in blood serum after 8-hour fasting.
Concentration of albumin | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of albumin in blood serum after 8-hour fasting.
Procalcitonin level | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of procalcitonin level (µg/L) in blood serum after 8-hour fasting.
White blood cells (WBC) count level | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  White blood cells (billion/L) count level in blood serum after 8-hour fasting
Lymphocyte count level | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Lymphocyte count (%) level in blood serum after 8-hour fasting
Platelet count level | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Platelet count level (billion/L) in blood serum after 8-hour fasting
Calculation of Nuclear index of intoxication (NII) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Calculated by dividing the number of myelocytes, young and stab neutrophils by number of segmented neutrophils.
Calculation of Leukocyte index of intoxication (LII) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Calculated by the formula of Kalf-Kalifa: correlation between the level of neutrophils and the content of other cells in the blood leukocytic composition.
Concentration of C-reactive protein (CRP) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of C-reactive protein (CRP) in blood serum after 8-hour fasting
Level of circulating immune complexes (CIC) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Level of Circulating immune complexes (CIC) in blood serum after 8-hour fasting
Concentration of Interleukin-1 and 2 | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of Interleukin-1 (pg/ml) and Interleukin-2 (pg/ml) in blood serum after 8-hour fasting
Calculation of neutrophil-to-lymphocyte ratio (NLR) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Calculated by dividing the number of neutrophils (%) by number of lymphocytes (%).
Concentration of immunoglobulins | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of Ig A, Ig M and Ig G in blood serum after 8-hour fasting
Concentration of complements | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Concentration of complements (C3, C4) in blood sample after 8-hour fasting
Assessment of central hemodynamics | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Measurement of central venous pressure (mmh2o) in the central vein
A change in the total Glasgow Coma Scale (GCS) score vs. baseline score upon admission | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  The GCS is composed of 3 components: ocular response (assessment 1-4 points), motor response (assessment 1-6 points) verbal response (evaluation of 1-5 points). Scores for each component are added together to get the total that will range between a minimum of 3 points (which corresponds to a patient who does not open his eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a patient with open eyes, obeying orders and maintaining a consistent language).
Assessment of electrocardiogram (ECG) | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Presence of clinically significant changes on ECG is evaluated.
Clinical signs | Will be evaluated for the duration of Intensive Care Unit (ICU) stay, at screening (Day 0) and Visit 3 (Day 3) of ICU stay.
  Presence of clinical signs (adynamia, weakness, memory impairment, sleep disorder, irritability) is based on patient's subjective complaints.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse events | Patients will be followed during 14 days.
  All types of adverse events
Incidence of multiple organ failure | Patients will be followed during 14 days.
  Incidence of multiple organ failure
Overall survival (%) at follow-up visit. | Follow-up visit (Day 14±1)
  Overall survival (%) at follow-up visit.

CONTACTS AND LOCATIONS:
Locations (13):
- Georgia (2):
  - "Unimedi Adjara" LLC, Batumi
  - Kutaisi Referral Hospital, Kutaisi
- Hospital of the Medical Center of the Administration of the President of the Republic of Kazakhstan, Astana, Kazakhstan
- Moldova (3):
  - Institute of Ambulance, Chisinau
  - Municipal Clinical Hospital "Sfinta Treime", Chisinau
  - Republican Clinical Hospital, Chisinau
- Ukraine (6):
  - Dnipro's Medical Academy of Ministry of Health of Ukraine, Dnipro
  - Zaicev's Institute of general and urgent surgery NMA Ukraine, Kharkiv
  - Khmelnytskyi Regional Clinical Hospital, Khmelnytskyi
  - HSEE of Ukraine "Ukrainian Medical Stomatological Academy"; Poltava Central District Hospital, Poltava
  - Central District Clinical Hospital, Vinnitsa
  - Zaporizka Medical Academy of postgraduate education, Zaporizkyi Clinical Hospital N9, Zaporizhzhya
- Republic Centre of Ambulance, Tashkent, Uzbekistan